CLINICAL TRIAL: NCT04034381
Title: Dietary Intake, Health and Micronutrient Status in Haiti: Establishing a Baseline to Manage and Evaluate a National Food Fortification Program
Brief Title: Dietary Intake, Health and Micronutrient Status in Haiti
Status: Terminated | Type: Observational
Why Stopped: Study suspended due to civil unrest and corresponding safety concerns and logistical challenges.
Sponsor: University of California, Davis (Other)
Collaborators: Le Ministère de la Santé Publique et de la Population, Haiti (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Global Alliance for Improved Nutrition (Other); Partners of the Americas (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1284500; 1718-68 (Other: Comité National de Bioéthique, Haiti)
Record Dates: First submitted 2019-02-27; First posted 2019-07-26 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Micronutrient Deficiency; Malnutrition, Child; Malnutrition; Chronic Disease
Keywords: Micronutrient deficiency; Dietary intake; Food fortification; National survey
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition; Chronic Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Port-au-Prince metropolitan area
  Interventions: Other: No intervention (descriptive survey only)
- Other urban areas
  Interventions: Other: No intervention (descriptive survey only)
- Rural areas
  Interventions: Other: No intervention (descriptive survey only)

INTERVENTIONS:
Other: No intervention (descriptive survey only) — No intervention

SUMMARY:
The general objective of this project is to collect information on dietary intake and nutritional status of women and young children in Haiti, to inform the design and management of national and subnational micronutrient intervention programs, with a focus on large-scale food fortification, and to serve as a reference point for program evaluation.

DETAILED DESCRIPTION:
Women of reproductive age and young children are especially vulnerable to micronutrient deficiencies which may lead to life-long disabilities. In Haiti, deficiencies in micronutrients such as iron, zinc, and vitamin A, are likely prevalent, but recent national estimates of the burden are not available. The most recent Demographic and Health Survey reported that 49% of women of reproductive age and 66% of preschool children were anemic. In addition, the Haitian population also has a high prevalence of overweight and obesity, with 38.5% classified as either overweight or obese. Fortification of staple foods with micronutrients is considered a cost-effective intervention to reduce the burden of micronutrient deficiencies. Through the Copenhagen Consensus Haiti Priorise exercise, fortification of flour with iron and folic acid was identified as the Number 2 development priority for Haiti. Prior to implementing a large-scale fortification program, however, the World Health Organization recommends the collection of detailed baseline information on nutritional status and dietary intake in the target population. In addition, information on certain biochemical indicators of nutritional status is needed to confirm the need for program implementation and to establish a baseline for later program evaluation and modification. Data on dietary patterns and nutrient intake are needed to 1) adapt nutrition intervention programs to match dietary nutrient gaps, and 2) design and manage complementary programs to address nutritional deficiencies in at-risk population subgroups that may not be reached or effectively covered by large-scale fortification programs.

The general objective of this project is to collect information on dietary intake and nutritional status of women and young children in Haiti, to inform the design and management of national and subnational micronutrient intervention programs, with a focus on large-scale food fortification, and to serve as a reference point for later program evaluation.

The specific objectives of the project are:

1. To describe the prevalence, at national and subnational levels, of anemia and selected micronutrient deficiencies among women and young children in Haiti (in addition to health indicators such as systemic inflammation, malaria infection, and anthropometric indices), to serve as a reference point for management and evaluation of a large-scale food fortification program, and other nutrition-related programs.
2. To measure dietary intake of micronutrients and potentially fortifiable foods, using 24-hour dietary recalls and the Fortification Assessment Coverage Toolkit (FACT), to confirm appropriate food vehicles for fortification, and to determine the specific micronutrients and fortification levels to be included in the program.
3. To measure micronutrient content in wheat flour samples collected from households, markets and/or bakeries to assess the current reach and fortification levels of fortified wheat flour.
4. To collect information on access to and use of public and private health care services and government programs (including food aid), to identify platforms, and their associated costs, for delivering nutrition programs to individuals not reached by large-scale food fortification.
5. To assess biological and behavioral risk factors for noncommunicable diseases, including blood glucose and lipid levels, to identify associations with health and nutritional status among women.
6. To measure micronutrient concentrations in human milk to assess micronutrient status of mothers and micronutrient intake of breastfeeding children.
7. To collect images to assist in the development of a novel digital anthropometric assessment method (technology for measurement of body size using photos).

The study will be designed as a stratified cluster survey with three ecological strata. Enumeration areas (clusters) and households within each cluster will be selected such that the sample is representative at the stratum level and national level.

ELIGIBILITY:
Inclusion Criteria:

* There is at least one child 6-59 months of age (the index child) in the household
* The primary or secondary female caregiver of the child who is 15-49 years of age (the index caregiver) is present in the household

Exclusion Criteria:

* The index child or index caregiver has fever, diarrhea with dehydration, or another serious health problem, or had any one of these conditions beginning on the day before the eligibility interview.

In addition, any lactating woman in the household is eligible for inclusion in the human milk assessment if she is breastfeeding an infant that is at least 30 days old. The lactating woman will be excluded from participating in the human milk assessment if she has a fever, diarrhea with dehydration, or another serious health problem, or had any of these conditions beginning on the day before the eligibility interview.

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be designed as a stratified cluster survey with 3 ecological strata. Enumeration areas (clusters) and households within each cluster will be selected such that the sample is representative at the stratum level and national level. The study will include households in which there is a child 6-59 months of age and a woman 15-49 years of age who serves as the child's primary caregiver.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2019-01-26 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Household-level consumption of "fortifiable" foods | Previous 7 days
  Measured using the Fortification Assessment Coverage Toolkit
Individual consumption of "fortifiable" foods | Previous 24 hours
  Assessed using repeated 24-hour dietary recalls
Vitamin A status among women and children | Single time point (1 day)
  Retinol in plasma or breast milk, and retinol-binding protein in plasma (micromol/L)
Zinc status among women and children | Single time point (1 day)
  Plasma zinc concentration (micrograms per dL)
Iron status among women and children | Single time point (1 day)
  Plasma ferritin concentrations (micrograms per L)
Folate status among women | Single time point (1 day)
  Red blood cell folate concentrations (nmol/L)
Vitamin B12 status among women and children | Single time point (1 day)
  Plasma vitamin B12 concentrations (pmol/L)
Micronutrient content of wheat flour samples collected from markets and bakeries | Single time point (1 day)
  Concentration of iron and zinc in wheat flour samples (mg/kg)
Usual nutrient intakes among women and children | 30 days (Previous month)
  Estimated population usual intakes of energy, fat, protein, carbohydrate, vitamin A, iron, zinc, folate, vitamin B12, thiamin, riboflavin, and niacin (based on combined data from 24-h dietary recalls and 30-day supplement questionnaire)

SECONDARY OUTCOMES:
Body mass index among women | Single time point (1 day)
  Body mass index, calculated as kg/m^2
Mid-upper arm circumference among children | Single time point (1 day)
  Mid-upper arm circumference, measured in mm
Height-for-age Z-score among children | Single time point (1 day)
  Height-for-age Z-score calculated using the WHO Growth Standard
Weight-for-age Z-score among children | Single time point (1 day)
  Weight-for-age Z-score calculated using the WHO Growth Standard
Weight-for-length Z-score among children | Single time point (1 day)
  Weight-for-length Z-score calculated using the WHO Growth Standard
Prevalence of malnutrition among children | Single time point (1 day)
  Prevalence of height-for-age, weight-for-age, or weight-for-height Z-score below <-2SD
Glucose concentration | Single time point (1 day)
  Glucose concentration in whole blood
Concentration of total cholesterol | Single time point (1 day)
  Concentration of total cholesterol in whole blood, mg/dL
Hemoglobin A1C concentrations | Single time point (1 day)
  Hemoglobin A1C concentrations in whole blood
Concentration of HDL cholesterol | Single time point (1 day)
  Concentration of HDL cholesterol in whole blood, mg/dL
Concentration of triglycerides | Single time point (1 day)
  Concentration of triglycerides in whole blood, mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Joseline Marhone Pierre, PhD, Study Chair — Ministère de la Sante Publique et de la Population, Haiti; Reina Engle-Stone, PhD, Principal Investigator — University of California, Davis; Stephen A Vosti, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Partners of the Americas, Pétionville, Haiti

IPD SHARING:
Plan to Share IPD: No